CLINICAL TRIAL: NCT05853640
Title: Patients With Longstanding HIP and Groin Pain Referred to Orthopedic Care: Effectiveness of Education and exerciSe ThERapy (HIPSTER)
Brief Title: Education and Exercise for Patients With Longstanding Hip and Groin Pain
Acronym: HIPSTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-05023-01
Record Dates: First submitted 2023-02-22; First posted 2023-05-11 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hip Pain Chronic; Femoro Acetabular Impingement; Groin Injury
Keywords: Hip-related pain; Longstanding hip and groin pain; Exercise therapy; Rehabilitation
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: 1:1 double blind randomized controlled trial, conforming to the CONSORT statement
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessors, and participants will be blinded to group allocation. An independent statistician, blinded to treatment allocation, will perform the statistical analysis. Treatment providers will be blinded to study hypothesis and the content of the different treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Participants in this group will undergo usual care at the orthopedic department and will get a recommendation for physical therapist-led treatment in primary care.
  Interventions: Other: Usual care
- HIPSTER (Experimental): Participants in this group will undergo usual care at the orthopedic department and will also receive a semi-structured intervention according to the HIPSTER treatment model.
  Interventions: Other: HIPSTER

INTERVENTIONS:
Other: Usual care — Usual care at the orthopedic department consists of a clinical examination, radiological imaging, and a diagnostic injection. A recommendation to get physical therapy treatment in primary care will be provided, but this intervention will not be controlled by the investigators in any capacity.
  Arms: Usual care
Other: HIPSTER — Patients will be provided with usual care at the orthopedic department, which consists of a clinical examination, radiological imaging, and a diagnostic injection.
  In addition, participants in this group will be referred to physical therapists trained in administering a semi-structured, individualized, progressive treatment. This 16-week intervention targets known physical and psychological impairments in people with long-standing hip and groin pain, using exercise therapy and patient education.
  Arms: HIPSTER

SUMMARY:
Longstanding hip and groin pain (LHGP) is a common and debilitating problem in young to middle aged individuals. These patients often get referred to orthopedic departments. Consensus statements on the management of these patients commonly recommend a physical therapist-led intervention as the first line intervention. However, the optimal content and delivery of this intervention is currently unknown. In this study we will compare the effectiveness of usual care (unstructured physical therapist-led intervention) to a semi-structured, progressive individualized physical therapist-led intervention on hip-related quality of life in people with longstanding hip and groin pain referred to an orthopedic department.

DETAILED DESCRIPTION:
This study is a parallel-group randomized controlled trial, comparing the effectiveness of patient education and exercise therapy to usual care on hip-related quality of life in people with longstanding hip and groin pain referred to an orthopedic department. Participants will be allocated in a 1:1 ratio to either usual care (orthopedic diagnostic pathway and recommendation of physical therapy) or the HIPSTER model, a semi-structured, progressive and individualized physical therapist-led intervention focusing on patient education and exercise therapy.

The primary aim of this trial is to determine the effectiveness of a structured physical therapist-led treatment model (HIPSTER) compared to usual care on hip-related quality of life. The primary hypothesis is that the HIPSTER model will be superior to usual care by at least 10 points between group change in improving self-reported hip-related function and quality of life, measured by iHOT-33.

Secondary aims include comparing group differences in achievement of patient acceptable symptom state (PASS) at 4 months and to compare between group changes in self-reported physical activity, pain self-efficacy, and pain catastrophizing, and physical performance tests regarding ROM, muscle force production, hop performance and balance between the HIPSTER group and usual care (baseline to 4 months), as well as cost-effectiveness of the interventions.

A full trial protocol will be published. The primary analysis will be performed using a t-test, according to intention-to-treat principles. A per protocol analysis will also be conducted, comparing participants who completed usual care or the HIPSTER model with high fidelity. Relevant parametric and non-parametric tests will be performed to compare change in physical performance tests and secondary PROMs.

A subgroup of patients will be included in qualitative study, using a semi-structured interview to capture the experience of participating in the HIPSTER intervention. Another subgroup will perform more advanced biomechanical analysis, including 3d-motion analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-55 years
* Referred to the Dept of Orthopedics due to hip and/or groin pain
* Activity-related unilateral or bilateral groin pain >3 months
* Pain reproduced with the FADIR test.

Exclusion Criteria:

* Groin pain originating from any diagnosis with other treatment pathways, i.e., i) Acute traumatic hip injuries (such as hip dislocation, hip fractures); ii) Verified moderate or severe OA (Tönnis grade >1); iii) Palpable hernia; iv) Low-back pain with a positive straight leg raise test and/or hip and groin pain provoked primarily by repeated motions of the lumbar spine; v) Sacroiliac joint pain with thigh thrust test.
* Co-morbidities potentially interfering with treatment, i.e., i) Co-morbidities overriding the hip and groin-related symptoms and dysfunction (such as other acute lower limb injuries, rheumatoid arthritis etc), ii) Co-morbidities prohibiting physical activity and training (heart disease etc), iii) Current psycho-social disorders requiring treatment.
* Other: i) History of drug abuse within the last year; ii) Not understanding the language of interest (Scandinavian languages, or English).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in iHOT-33 scores at 4 months | The primary outcome will be collected at baseline and at the primary end-point (4 months after baseline).
  iHOT-33 is a 33 question self-reported outcome scale, measuring hip-related quality of life. This outcome measure has been validated and translated to Swedish. The scores are summed on a 0 (worst)-100 (best) scale.

SECONDARY OUTCOMES:
Change in iHOT-33 scores at 1, 2 and 5 years | This outcome will be collected at baseline and 1,2 and 5 years after baseline.
  iHOT-33 is a 33 question self-reported outcome scale, measuring hip-related quality of life. This outcome measure has been validated and translated to Swedish. The scores are summed on a 0 (worst)-100 (best) scale.
Patient acceptable symptom state (PASS) | This outcome will be collected at the primary endpoint (4 months after baseline). In addition it will also be collected at 1,2 and 5 years after baseline.
  The patient acceptable symptom state (PASS) will be collected using a dichotomized question ("Taking into account your hip and groin function and pain, and how it affects your daily life, including your ability to participate in sport and social activities, do you consider that your current state is acceptable if it remained like that for the rest of your life?").
Treatment failure | This outcome will be collected at the primary endpoint (4 months after baseline). In addition it will also be collected at 1,2 and 5 years after baseline.
  Treatment failure will be collected using a dichotomized question "Do you consider your current state so unsatisfactory that you think your treatment has failed?".
Perceived symptom improvement | This outcome will be collected at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Perceived symptom improvement will be collected using a 7-point Global rating of change (GROC) scale, ranging from -3 (a lot worse), to +3 (a lot better).
Patient desire and beliefs regarding surgical intervention | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Patient desire and beliefs regarding surgical intervention will be collected using two dichotomized questions; "Do you want to undergo surgery?" and "Do you believe surgery is needed for you to get better?".
Physical activity | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Physical activity and return to sport/exercise will be collected using questions based on the Swedish National Board of Health and Welfare (Socialstyrelsen) physical activity screening, a self-reported measure of minutes spent doing strenuous and everyday activities.
Pain catastrophizing | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Pain catastrophizing will be measured with the Pain Catastrophizing Scale (PCS), a valid patient-reported outcome with 13 items. It is scored 0 to 52, with higher values indicating higher degrees of catastrophizing.
Pain self-efficacy | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Pain-related self-efficacy will be collected with the short-form Pain Self-efficacy Questionnaire (PSEQ-2), a commonly used measure of self-efficacy in musculoskeletal pain. PSEQ-2 consists of 2 questions. It is scored 0 to 12, with higher score indicating a greater degree of pain self-efficacy.
Health related quality of life | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Generic health-related quality of life will be measured using EQ5D. It is scored from 0 to 1, where 1 corresponds to perfect health, and is available in Swedish.
Employment status | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Employment status will be measured using a Likert scale, from unemployed, student, part time work, full time work or retired.
Surgical interventions | This outcome will be collected from medical records at 1, 2 and 5 years.
  Any performed surgical interventions to the hip and/or groin region will be collected from medical records and self-reported questions.
Osteoarthritis development | This measure will be collected at baseline, and at 2 and 5 year follow ups.
  The presence of narrowing joint space will be measured using Tönnis grade, measured on an AP radiograph.
Usual care content | This outcome will be collected from the usual care group, after the primary end-point at 4 months.
  Any physical therapist-led intervention in the usual care group will be collected using self-reported questions regarding volume (number of sessions), content (overall focus of intervention) and adherence (patient compliance to prescribed intervention).
Hip range of motion | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Hip range of motion (in degrees) will be measured with a digital inclinometer in internal rotation in 90° of hip flexion and zero° flexion.
Isometric hip muscle force production | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Isometric hip muscle force production will be measured (in Newton and nm/kg) with a belt-fixated handheld dynamometer for hip adduction, flexion and hip extension.
Hop performance | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Hop performance will be assessed using the single leg hop for distance test. Distance (cm) and kinematics (joint angles) and forces (joint moments) will be measured.
Y-balance test | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Single leg balance will be assessed using the Y-balance test. Distance (cm) and Limb symmetry index will be collected.
Single leg balance | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Single leg balance will be evaluated by postural sway using markers, 3D-motion capture and force plates.
Single leg squat | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Single leg squat performance will be evaluated using markers, 3D-motion capture and force plates to calculate kinematics (joint angles) and kinetics (joint moments) related to the task.
Step down | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Step down performance will be evaluated using markers, 3D-motion capture and force plates to calculate kinematics (joint angles) and kinetics (joint moments) related to the task.
Rear foot elevated split squat jump | This outcome will be collected at baseline and at the primary endpoint (4 months after baseline). In addition it will also be collected at 1 year after baseline.
  Lower body power will be evaluated using markers, 3D-motion capture and force plats to collect kinematics (joint angles) and kinetics (joint moments) during the task.

OTHER OUTCOMES:
Qualitative interviews - Patients | The interviews will be conducted between 4 months and 6 months after baseline.
  A sub-group of participants (about 10 or until saturation) will be interviewed in a semi-standardised fashion, about their experiences of undergoing the intervention.
Qualitative interviews - Physical therapists | The interviews will be conducted during active data collection, when clinicians have treated a minimum of 3 patients in the trial, with an estimated average of 6 months after data collection has started.
  Physical therapists trained in delivering the intervention in the experimental arm will be interviewed in a semi-standardised fashion, about their experiences of treating this patient population and their experience of delivering the experimental intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Lund University
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to Swedish laws and regulations, individual data points cannot be shared.